CLINICAL TRIAL: NCT05762380
Title: In Vitro Fecal Fermentation Following Ingestion of Iron-enriched Aspergillus Oryzae or Iron Sulfate
Brief Title: Effect of Iron Supplements on the Growth of Enteric Pathogens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor Doris A. Adams Endowed Chair, Iowa State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IVFE
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-09

CONDITIONS: Iron-deficiency; Iron Deficiency Anaemia Due to Dietary Causes; Iron Deficiency Anemia Treatment; Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: FeSO4 Dietary Supplement: Ao iron
Who Masked: Participant, Investigator
Masking Description: This is a double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferrous sulfate (FeSO4) (Active Comparator): FeSO4 supplements containing 54 mg elemental iron
  Interventions: Dietary Supplement: Ferrous sulfate
- Ferrous sulfate-enriched Aspergillus oryzae (Ao iron) (Experimental): Ao iron supplements containing 54 mg elemental iron
  Interventions: Dietary Supplement: Ferrous sulfate-enriched Aspergillus oryzae (Ao iron)

INTERVENTIONS:
Dietary Supplement: Ferrous sulfate — 2 FeSO4 supplements containing 27 mg elemental iron/supplements (54 mg total iron)
  Arms: Ferrous sulfate (FeSO4)
Dietary Supplement: Ferrous sulfate-enriched Aspergillus oryzae (Ao iron) — 2 Ao iron supplements containing 27 mg elemental iron/supplements (54 mg total iron)
  Arms: Ferrous sulfate-enriched Aspergillus oryzae (Ao iron)

SUMMARY:
Iron supplementation is a common approach to address iron deficiency with recommendations for women of childbearing age, particularly those at risk of iron deficiency. Because of its considerably higher absorption, ferrous sulphate is the common iron compound used in iron supplements. However, concerns about iron supplements arise from the knowledge that a large portion of the supplement consumed is not absorbed. This unabsorbed iron travels to the colon and, in preclinical studies, has been shown to promote the growth of enteric pathogens at the expense of beneficial commensal bacteria and increase infection risk, including the clinical incidence of diarrhea. The objective of this study is to compare the effects of iron as ferrous sulfate (FeSO4) or FeSO4-enriched Aspergillus oryzae (Ao iron) on the growth and virulence of common enteric pathogens using an in vitro fecal fermentation model. Stool samples will be collected from women of reproductive age following ingestion of an iron supplement as either FeSO4 or Ao iron. Stool samples will be spiked with common enteric pathogens, and outcome measures will be determined following in vitro fecal fermentation.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-44 y
* Are able to swallow the iron pills provided for the study
* BMI 18.5 to 29.9 kg/m2
* Willing to provide blood samples
* Willing to collect stool samples

Exclusion Criteria:

* Currently taking any antibiotics
* Iron overload condition/hemochromatosis
* History of chronic gastrointestinal disorders/diseases
* Currently smoke cigarettes (including vaping)
* Have donated blood recently (in the last two weeks)
* Currently taking a vitamin and mineral supplement containing iron
* Pregnant and lactating/breastfeeding women
* Allergic to any of the ingredients (wheat, egg, butter, milk, and baking powder, blue dye) in the muffins

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation of gender identity at birth
Enrollment: 15 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Concentration of iron taken up by enteric pathogens | Time Frame: 0-24 hours
  Iron uptake of common enteric pathogens will be determined in stool following in vitro fecal fermentation.
Growth of enteric pathogens measured by optical density | Time Frame: 0-24 hours
  Growth of common enteric pathogens will be determined in stool following in vitro fecal fermentation.

SECONDARY OUTCOMES:
Gut microbiome composition and diversity | Time Frame: 0-24 hours
  Gut microbiome composition will be determined in stool following in vitro fecal fermentation using 16S rRNA gene sequencing.
Individual fecal short chain fatty acid (SCFA) concentration | Time Frame: 0-24 hours
  Individual SCFAs will be determined in stool following in vitro fecal fermentation by liquid chromatography-mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, Ph.D., Principal Investigator — Iowa State University
Locations (1):
- Iowa State University, Ames, Iowa, United States